CLINICAL TRIAL: NCT05745194
Title: Nutritional Counselling Promoting Adherence to the Mediterranean Diet as Adjuvant in the Treatment of Major Depressive Disorder: A Randomized Open Controlled Trial Study
Brief Title: Influence of Nutrition in Depression Treatment (INDEPT)
Acronym: INDEPT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Associacao para Investigacao e Desenvolvimento da Faculdade de Medicina - CETERA (Other)
Collaborators: University of Lisbon (Other); Instituto Politécnico de Leiria (Other); Fundação para a Ciência e a Tecnologia (Other)
Responsible Party: Principal Investigator, Maria João Heitor, Head of Psychiatry, Principal Investigator, Associacao para Investigacao e Desenvolvimento da Faculdade de Medicina - CETERA
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PTDC/SAU-NUT/3321/2020
Record Dates: First submitted 2023-01-25; First posted 2023-02-27 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Major Depressive Disorder - MDD
Keywords: Depression; Major Depressive Disorder; Nutritional Intervention; Randomized Controlled Trial; Mediterranean Diet
MeSH Terms: conditions — Depression; Depressive Disorder, Major

STUDY DESIGN:
Intervention Model Description: The study will follow a randomized open controlled trial design with concealment of participants allocation to the researchers involved in data collection at the end of the trial and follow-up assessments.
  Researchers participating in the statistical analysis of the trial´s data will also be concealed to group allocation.
  Participants meeting all inclusion criteria will be randomized to (a) the intervention group: six nutritional consultations with a registered nutritionist promoting adherence to the MedDiet and TAU or (b) the control group: only exposed to TAU for MDD.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The researchers responsible for the data collection at the end of the trial and follow up assessments will be hired and trained by the study staff exclusively for that task to mitigate potential bias.
  The statistical analysis will be performed by researchers, prior to the unblinding of participants. The unmasking of participants group allocation will only occur after the statistical analysis of the clinical trial results at 12-week is performed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional Group (Experimental): Interventional group with six nutritional counselling consultations promoting the adherence to the MedDiet and TAU for MDD
  Interventions: Behavioral: Promotion of adherence to the MedDiet
- Control Group (No Intervention): Individuals with TAU for MDD

INTERVENTIONS:
Behavioral: Promotion of adherence to the MedDiet — Participants will be followed in six individual nutrition consultations with a duration of 30 to 60 minutes. The consultations will be focused on promoting the adherence to the MedDiet.
  The nutritional intervention will be personalized to each individual ad libitum, without calories or macronutrients restriction and without the goal to promote weight change. The intervention will begin with an initial assessment of the dietary patterns of the participants in which the nutritionist will identify potential behavioural changes to promote adjustments in dietary habits and therefore adherence to the MedDiet.
  The intervention will promote positive recommendations (behaviours recommended to follow) and negative recommendations (behaviours recommended to reduce or eliminate) (26), using the strategy and MedDiet definition proposed by Estruch et al. in the "Primary Prevention of Cardiovascular Disease with a Mediterranean Diet" study (3).
  The participants will also maintain MDD TAU.
  Arms: Interventional Group

SUMMARY:
The hypothesis to be tested by this study is that an intervention promoting adherence to the MedDiet can decrease symptoms of depression in patients with elevated inflammation biomarkers, namely C-reactive protein (CRP) and Interleukin 6 (IL-6) diagnosed with Major Depression Disorder (MDD), under treatment with antidepressant medication for a period of time less than or equal to 6 months.

The main aim of this study is to understand if promoting the adherence to the MedDiet, as an adjuvant strategy in the treatment of MDD, is effective in decreasing symptoms of depression in MDD patients, with elevated levels of inflammation biomarkers.

Other specific objectives of the study are

1. To assess the association between adherence to MedDiet and changes in inflammatory biomarkers;
2. To assess the association between changes in inflammatory biomarkers with symptoms of MDD;
3. To evaluate the association between adherence to MedDiet and effectiveness of psychiatric treatment of MDD;
4. To characterize the association between adherence to MedDiet and changes in health-related quality of life
5. To evaluate the economic cost-effectiveness of dietary counselling, as an adjuvant treatment in MDD.

The study will have a duration of 12 weeks, with a randomized parallel-group open controlled trial design, with two parallel groups with an allocation ratio of 1:1 - (a) intervention arm with six nutritional consultations with a registered nutritionist, promoting adherence to MedDiet, in addition to MDD Treatment-As-Usual (TAU) and (b) control group arm benefitting only from MDD TAU. A follow up assessment will be performed at 6- and 12-months.

Having into consideration an attrition of 40 percentage at the end of the intervention, the minimum sample size estimated is 190 (95 per arm).

The main outcome of the trial, changes in symptoms of depression, will be evaluated using the Beck Depression Inventory Second Edition (BDI-II).

DETAILED DESCRIPTION:
To test the study´s hypothesis, namely if an intervention promoting adherence to the MedDiet can decrease symptoms of depression in patients with MDD and elevated inflammation biomarkers, the following objectives will be assessed.

The main objective of the trial is:

1.To assess the effectiveness of dietary counselling promoting MedDiet, as an adjuvant treatment of MDD, to decrease depressive symptoms in adults diagnosed with MDD and having elevated inflammation biomarkers (CRP, IL-6).

Specific objectives are:

1. To assess the association between adherence to MedDiet and changes in inflammatory biomarkers
2. To assess the association between changes in inflammatory biomarkers with symptoms of MDD
3. To evaluate the association between adherence to MedDiet and effectiveness of psychiatric treatment of MDD
4. Characterize the association between adherence to MedDiet and changes in health-related quality of life
5. To evaluate the economic cost-effectiveness of dietary counselling, as an adjuvant treatment in MDD

This study is a 12-week multicentre randomized parallel-group open controlled trial, with a follow up assessment at 6- and 12-months after baseline data collection, with two parallel groups with an allocation ratio of 1:1. - (a) intervention arm with six nutrition consultations with a registered nutritionist, promoting adherence to MedDiet, in addition to MDD treatment as usual (TAU) and (b) control group benefitting only from MDD TAU. Participants will be individuals diagnosed with a first episode of MDD, according to the "F32 Depressive episode" (F32.0; F32.1; F32.2) classification of the Tenth Revision of the International Classification of Diseases (ICD-10), under treatment with antidepressant medication for a period of time less than or equal to 6 months, attending to outpatient consultations.

Potential participants will be invited to enrol by their medical doctors from the participating recruitment centres. The invitation will be made at regular medical appointments including primary care consultations and outpatient psychiatric consultations in one of the participant centers. After signing the informed consent, CRP and IL-6 levels will be tested. Participants with increased inflammatory biomarkers, meeting all other inclusion criteria will be randomized to (a) the intervention arm or (b) the control arm of the study, in a 1:1 ratio, using a computer-generated list of random numbers stratified by center in variable blocks of size 2, 4 and 6. Treatment allocation will be concealed from the researchers, using sequentially numbered, opaque, sealed envelopes.

The study will use a convenience sample from patients diagnosed with MDD attending to outpatient consultations in one for the participating clinics.

Considering a 2-sided significance level of 5 percent and a power of 80 percent and having into consideration an attrition of 40 percent at the end of the intervention, the minimum sample size estimated is 190 (95 per arm). Estimating a prevalence of elevated inflammation in 30 percentage of MDD patients and 10 percentage of patients that don't meet other inclusion criteria, the number of recruited participants estimated is 700.

Participants allocated to the intervention group will attend six nutrition consultations, performed by a register nutritionist in weeks 1, 2, 4, 6, 8 and 10. The intervention will be personalized to each participant and will promote adherence to the Mediterranean Diet, ad libitum, without calories or macronutrients restriction or recommendation for weight change.

The intervention will follow a similar approach to the one proposed by Estruch et al. in the "Primary Prevention of Cardiovascular Disease with a Mediterranean Diet" study.

The intervention will contemplate the following recommendations:

Positive recommendations (promotion of the intake of the following foods):

1. Use of olive oil as main fat, both for cooking and dressing;
2. 2 or more servings of vegetables daily (200g of vegetables per serving);
3. 2-3 servings of fresh fruits per day;
4. 3 or more servings of legumes per day;
5. 3 or more servings of fish per week (100 - 150g of fish per serving or 200g of shellfish);
6. 3 or more servings of nuts a week (30g of nuts per serving);
7. Meat consumption mainly from poultry (without skin) or rabbit;
8. Home cooked meals with tomato, garlic and onion, at least twice a week;

Negative recommendations (eliminate or drastically reduce the following foods):

1. Cream, butter and margarine;
2. Cold meats, paté and duck meat;
3. Carbonated and/or sugared beverages;
4. Pastries and industrial baked products (cakes, donuts or cookies);
5. Industrial deserts;
6. French fries and potato chips;
7. Pre-cooked cakes and sweets;
8. If alcohol is consumed should be limited to 300ml of wine per day (150cc at meals for men and 100cc for woman, during meals);

Training of the nutritionists delivering the intervention will be provided prior to the beginning of recruitment and during the duration of the trial in MDD, therapeutic relationship, trauma and Mediterranean Diet.

Data analysis and reporting will be performed in accordance with Consolidated Standards of Reporting Trials (CONSORT) guidelines.

Primary analysis will include all randomized participants, following an intention-to-treat (ITT) approach. Baseline characteristics of the participants, by group, will be reported using descriptive statistics and compared by χ^2 and t-test for independent samples (or equivalent non-parametric test).

To evaluate the effectiveness of nutritional counselling promoting MedDiet, the scale BDI-II will be used categorically in accordance with the standardized cutoffs: minimal depression (0-13), mild depression (14-19), moderate depression (20-28), severe depression (29-63). The success measure will be a decrease in category in the severity of depressive symptoms. The proportion of participants with a decrease in depression severity symptoms category according to the BDI-II (main outcome) will be compared between control and intervention groups using generalized linear mixed models.

Further adjustment for relevant covariates, as supportive analysis, will be made. Secondary analyses, including the analysis of the main outcome measure (BDI-II) as a continuous variable, will be conducted using (Generalized) Linear Mixed Models, as appropriate. For each outcome, results for either intervention and control group, and estimates of effect size with a 95 percent confidence interval will be reported. All analyses will be performed using R and R Studio version 3.5.3 and R Studio version 1.3.618 (or another updated version in the moment of analysis), assuming a significance level of 5 percent.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 18-70 years old
2. Able to understand and provide informed consent
3. Able to read and write
4. Have a diagnosis of MDD (according to ICD-10 F32.0; F32.1; F32.2; F32.9; F33.0; F33.1; F33.2; F33.9 criteria)
5. Score on the Beck Depression Inventory-II scale (BDI-II) > 13;
6. Elevated biomarkers of inflammation (CRP > 3mg/l or IL-6 ≥ 2pg/ml )
7. Able to follow a MedDiet without impeditive physical or religious limitations, allergies or intolerances
8. Being under pharmacological treatment for depressive disorder

Exclusion Criteria:

1. Diagnosis of autoimmune diseases, thyroid dysfunction or cancer
2. Diagnosis of bipolar disorder, psychotic disorders, eating disorders
3. Self-reported acute infection 2 weeks prior to the blood sample collection
4. Pregnancy or lactation
5. Glucocorticoid medication
6. Prescribed with NMDA Receptor Antagonists
7. Under treatment with brain stimulation techniques for the depressive episode
8. Currently participating in another intervention targeting diet, physical exercise, or MDD treatment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2023-06-05 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in symptoms of MDD | Baseline, 12-weeks, 6-months, and 12-months after the baseline assessment
  Symptoms of depression will be assessed with the self-administered Beck Depression Inventory-II (BDI-II) scale. To measure changes in the main outcome, the score of the BDI-II will be used categorically, considering the cut-offs proposed: 0-13 minimal depression; 14-19 mild depression; 20-28 moderate depression; 29-63 severe depression. The success measure will be a downgrade of category in the severity of depressive symptoms. The analysis of the score of the BDI-II will also be performed using the scale score as a continuous variable.

SECONDARY OUTCOMES:
Inflammation biomarkers (IL-6 and/or CRP) | Baseline, 12-weeks, 6-months, and 12-months after the baseline assessment
  Identification of statistically significant variation of IL-6 and/or CRP concentrations in blood between baseline and other moments of assessment.
  CRP and IL-6 will be measured using a Atellica CH Analyzer.

OTHER OUTCOMES:
Adherence to the Mediterranean Diet according to the 14-point Mediterranean Diet Adherence Screener Scale | Baseline,12-weeks, 6-months, and 12-months after the baseline assessment
  The Adherence to the Mediterranean Diet will be assessed by the validated Portuguese version of the 14-point Mediterranean Diet Adherence Screener. This instrument evaluates the intake of foods typical of the MedDiet. The scale presents a result from 0 to 14 points, with a higher score indicating greater adherence to the mediterranean dietary pattern.
  Changes between baseline and other assessments will be analysed using the score of the scale as a continuous variable..
Health-related quality of life | Baseline, 12-week, 6-months, and 12-months after the baseline assessment
  Changes in health-related quality of life between baseline and other assessment moments will be accessed by the World Health Organization Quality of Life - Brief (WHOQOL-BREF). The global score of the scale ranges from 0 to 100 points, with a higher score indicating a higher quality of life.
Healthcare use cost | Baseline,12-weeks, 6-months, and 12-months after the baseline assessment
  The estimation cost of healthcare resource use will be assessed using: number of days of hospital admission, general care medical appointments and specialty medical appointments, sessions of massage and physiotherapy, psychology appointments and ocupational therapy appointments.
Absenteeism | Baseline,12-weeks, 6-months, and 12-months after the baseline assessment
  Absence from work will be estimated in hours.

CONTACTS AND LOCATIONS:
Overall Officials: Maria João Heitor, PhD, Principal Investigator — Instituto de Saúde Ambiental, Faculdade de Medicina da Universidade de Lisboa, Portugal
Locations (2):
- Portugal (2):
  - Hospital de Beatriz Ângelo - Hospital de Loures, EPE, Loures, Lisbon District
  - Centro Hospitalar de Leiria - Hospital Santo André, Leiria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yang C, Wardenaar KJ, Bosker FJ, Li J, Schoevers RA. Inflammatory markers and treatment outcome in treatment resistant depression: A systematic review. J Affect Disord. 2019 Oct 1;257:640-649. doi: 10.1016/j.jad.2019.07.045. Epub 2019 Jul 5. PMID 31357161
- [Background] Osimo EF, Baxter LJ, Lewis G, Jones PB, Khandaker GM. Prevalence of low-grade inflammation in depression: a systematic review and meta-analysis of CRP levels. Psychol Med. 2019 Sep;49(12):1958-1970. doi: 10.1017/S0033291719001454. Epub 2019 Jul 1. PMID 31258105
- [Background] Estruch R, Ros E, Salas-Salvado J, Covas MI, Corella D, Aros F, Gomez-Gracia E, Ruiz-Gutierrez V, Fiol M, Lapetra J, Lamuela-Raventos RM, Serra-Majem L, Pinto X, Basora J, Munoz MA, Sorli JV, Martinez JA, Martinez-Gonzalez MA; PREDIMED Study Investigators. Primary prevention of cardiovascular disease with a Mediterranean diet. N Engl J Med. 2013 Apr 4;368(14):1279-90. doi: 10.1056/NEJMoa1200303. Epub 2013 Feb 25. PMID 23432189 (Retraction: PMID 29897867 N Engl J Med. 2018 Jun 21;378(25):2441-2442)
- [Background] Beck AT, Steer RA, Ball R, Ranieri W. Comparison of Beck Depression Inventories -IA and -II in psychiatric outpatients. J Pers Assess. 1996 Dec;67(3):588-97. doi: 10.1207/s15327752jpa6703_13. PMID 8991972
- [Background] Garcia-Conesa MT, Philippou E, Pafilas C, Massaro M, Quarta S, Andrade V, Jorge R, Chervenkov M, Ivanova T, Dimitrova D, Maksimova V, Smilkov K, Ackova DG, Miloseva L, Ruskovska T, Deligiannidou GE, Kontogiorgis CA, Pinto P. Exploring the Validity of the 14-Item Mediterranean Diet Adherence Screener (MEDAS): A Cross-National Study in Seven European Countries around the Mediterranean Region. Nutrients. 2020 Sep 27;12(10):2960. doi: 10.3390/nu12102960. PMID 32992649
- [Background] Gregorio MJ, Rodrigues AM, Salvador C, Dias SS, de Sousa RD, Mendes JM, Coelho PS, Branco JC, Lopes C, Martinez-Gonzalez MA, Graca P, Canhao H. Validation of the Telephone-Administered Version of the Mediterranean Diet Adherence Screener (MEDAS) Questionnaire. Nutrients. 2020 May 22;12(5):1511. doi: 10.3390/nu12051511. PMID 32455971
- [Background] Development of the World Health Organization WHOQOL-BREF quality of life assessment. The WHOQOL Group. Psychol Med. 1998 May;28(3):551-8. doi: 10.1017/s0033291798006667. PMID 9626712